CLINICAL TRIAL: NCT02025387
Title: Physical Activity in Patients With Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kidong Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH_GO_034
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Women Who Underwent Midline Incision, Gynecological Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Patients will receive physical activity feedback and be encouraged to achieve the daily goals of physical activity
  Interventions: Behavioral: Physical activity feedback
- Control (Sham Comparator): Physical activity will be measured but not be informed to patients. She will receive usual care.
  Interventions: Behavioral: Usual care except physical activity measurement

INTERVENTIONS:
Behavioral: Physical activity feedback
  Arms: Experimental
Behavioral: Usual care except physical activity measurement
  Arms: Control

SUMMARY:
Examine whether the measurement and feedback of physical activity increase the physical activity in women who underwent midline incision, gynecological surgery

ELIGIBILITY:
Inclusion Criteria:

* Midline incision, gynecological surgery

Exclusion Criteria:

* Cannot ambulate
* Anticipated long term ICU care
* Cannot wear accelerometer
* Anticipated discharge before postoperative day 5

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Physical activity recovery rate | Postoperative day 4 and 5
  Baseline physical activity is measured before admission. Specifically, on presurgery day 3 and 4, patients wear accelerometer. The average physical activity of presurgery day 3 and 4 is calculated and be regarded as baseline physical activity.
  After surgery, the average physical activity of postoperative day 4 and 5 is calculated. The ratio of the average physical activity of postoperative day 4 and 5 versus baseline physical activity is estimated. The ratio is physical activity recovery rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea